CLINICAL TRIAL: NCT00702286
Title: Phase II Prospective Comparison Randomized Placebo Controlled Double Blind Study to Evaluate the Efficacy of the UroShieldTM Surface Acoustics Ultrasound Device for the Treatment of Patients With Percutaneous Nephrostomy
Brief Title: Evaluation of Surface Acoustics Ultrasound Device for the Treatment of Patients With Percutaneous Nephrostomy Catheters
Acronym: NV-US-04-001
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Nanovibronix (Industry)
Responsible Party: Yoram Siegel MD Head of endourolgy unit assaf harofeh MC, Assaf Harofeh MC
Other Study IDs: 75/08
Record Dates: First submitted 2008-06-17; First posted 2008-06-20 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-05

CONDITIONS: Urinary Tract Infection
Keywords: Surface acoustic ultrasound; biofilm formation; percoutaneous nephrostomy tube; Patients requiring per coetaneous drainage due to urinary; tract obstruction; To evaluate the efficacy of surface acoustic wave in; reducing pain and improving drainage
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: None Retained — urine culture
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Two arm, double blinded, comparative, randomized, placebo controlled (active:sham - 2:1) study
- 2: Two arm, double blinded, comparative, randomized, placebo controlled (active:sham - 2:1) study

SUMMARY:
Catheter associated urinary tract infection is one of the most common types of catheter acquired infections and adds greatly to patient morbidity, mortality and medical cost. Urinary catheters may readily acquire biofilms when inserted. The longer the catheter remains in place, the greater the tendency of these organisms to develop biofilms and result in urinary tract infections, which are difficult to treathe UroShield System is intended to prevent bacterial biofilm formation by means of the Active NanoShield technology it has developed. A number of scientific concepts and principles shown in prior studies have shown some promising results in the treatment of biofilm based sequele using ultrasound energy. The NanoShield technological basis of the UroShield System has taken these concepts to a level where acoustical waves in the ultrasound range can be created by low cost disposable actuators which actually create a physical coating on all of the surfaces of the catheter thereby interfering with the attachment of bacteria which is the initial step in biofilm formation.

DETAILED DESCRIPTION:
The UroShield™ System is comprised of 2 main components:· The Disposable UroShield Z-Patch - a disposable small lightweight patch that is attached to the PCN catheter, while its opposite side is attached directly to the patient's skin at the site of catheter entry. The patch has twofold function:

1. it receives energy and a signal from the UroShield Driver allowing it to generate the ultrasonic waves;
2. it acts as a fixation device for the PCN catheter.· The UroShield Driver - an external driver unit that is attached to the UroShield patch and contains batteries to power the system and electronics that control the patch unit

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring percoutaneous nephrostome
* First insertion

Exclusion Criteria:

* Blood coagulation disorders
* Trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients requiring percoutaneous nephrostome drainage for period for more then 4 weeks
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2008-08

PRIMARY OUTCOMES:
Reduction in pain and discomfort in patients with PCN catheters, improvement of catheter's patency. | 28 days for one subject overall 1 year

SECONDARY OUTCOMES:
Renal function improvement | 28 days per pateint overall 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yoram I Siegel, MD, Principal Investigator — Assaf Harofeh MC
Locations (1):
- Assaf Harofeh MC, Ẕerifin, Isarel, Israel